CLINICAL TRIAL: NCT03948555
Title: Magnetic Resonance Imaging (MRI) for Aortic Dissection to Visualise Inflammation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0688
Record Dates: First submitted 2019-05-07; First posted 2019-05-14 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Aortic Dissection; Aortic Diseases
MeSH Terms: conditions — Aortic Dissection; Aortic Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute aortic dissection: stable patients with confirmed diagnosis of acute AD.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI) using ultrasmall super paramagnetic iron oxides (USPIOs)
- Chronic aortic dissection: patients with diagnosis of chronic AD, being followed up in outpatient aortic clinic.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI) using ultrasmall super paramagnetic iron oxides (USPIOs)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) using ultrasmall super paramagnetic iron oxides (USPIOs) — All patients will undergo two MRI scans (one MRI scan pre-USPIO administration, and one MRI scan 24-36 hours following USPIO administration) and blood samples will be taken for future biomarker analysis.

SUMMARY:
The study is a single-centre, prospective, observational cross-sectional imaging study aimed to determine if macrophage-mediated inflammation can be visualised in the aorta of patients with aortic dissection (AD) using ultrasmall super paramagnetic iron oxides (USPIO)-enhanced magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Aortic dissection (AD) is a condition in which a disruption of the medial layer (in most cases provoked by a tear or an ulcer in the intima) results in separation of the aortic wall layers, with concomitant 'false lumen' formation and malperfusion of end organs.

The underlying mechanism of the condition has, until recently, remained unclear. The Pi of the present sutdy has shed light on a mechanism that shows that inflammation underlies the condition. The PI of the present study has showed that inflammation in the aorta is triggered by macrophage infiltration into the aortic wall in both pre-clinical models using animal models of the condition (murine) and in patient tissue samples obtained at time of surgery.

Macrophage infiltration into the aortic wall, as a result of activation of the cytokine, granulocyte-macrophage colony stimulating factor (GM-CSF), is the trigger for an inflammatory cascade that is presently understood to underlie the pathogenic mechanism of the condition

Non-invasive assessment of macrophage infiltration would prove that this pathogenic mechanism exists (proof-of-concept). Macrophage infiltration has been shown to be feasible by contrast-enhanced Magnetic Resonance Imaging (MRI) using ultrasmall super paramagnetic iron oxides (USPIOs).

The hypothesis of the present study is that macrophage-mediated inflammation can be visualised in the aorta of patients with AD using the USPIO-enhanced MRI technique, and use the present study to confirm this (proof-of-concept).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute or chronic aortic dissection (>2 week after initial intimal injury)
* Able and willing to comply with all study requirements.
* Age > 40 years (Patients under the age of 40 years will not be included as they may have a connective tissue disorder accounting for their condition)
* Able and willing to give informed consent
* An adequate understanding of written and verbal English

Exclusion Criteria:

* Past history of systemic iron overload or haemochromatosis
* Renal failure (estimated glomerular filtration rate < 30ml/min)
* Contraindication to MRI
* Known allergy to iron-containing compounds
* Participants who have participated in another research study involving an investigational product in the past 12 weeks.
* Female participants who are pregnant or lactating.
* Unwilling or unable to give informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute patients will be identified in cardiologic inward, after that patients have been discharged from the coronary care unit at Glenfield Hospital, Leicester. Chronic patients will be identified from the aortic outpatient clinic at Glenfield Hospital.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Visualisation of inflammation | Up to 36 hours
  To determine if macrophage-mediated inflammation can be visualised in the aorta of patients with aortic dissection using USPIO-enhanced MRI
Feasibility | Up to 36 hours
  To establish the feasibility of imaging macrophage-mediated inflammation in the aorta of patients with aortic dissection, using USPIO-enhanced MRI.

SECONDARY OUTCOMES:
Timing | Up to 36 hours
  To determine the timing of macrophage infiltration in aortic dissection (acute or chronic phase)
Localisation | Up to 36 hours
  To assess if macrophage mediated inflammation is localised to the site of dissection and the surrounding aorta or more widespread in the vasculature.

CONTACTS AND LOCATIONS:
Overall Officials: Toru Suzuki, MD, PhD, Study Chair — University of Leicester
Locations (2):
- United Kingdom (2):
  - University of Leicester, Leicester
  - University Hospitals of Leicester NHS Trust, Leicester

IPD SHARING:
Plan to Share IPD: No